CLINICAL TRIAL: NCT06512857
Title: The Effect of Hand Puppets and Kaleidoscope on Pain and Fear in Preschool Children Who Had Skin Prick Tests in the Pediatric Allergy and Immunology Polyclinic
Brief Title: The Effect of Hand Puppets and Kaleidoscope on Pain and Fear in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Özlem Selime MERTER, ASSISTANT PROFESSOR, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/04-34
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Nursing Caries; Pain; Fear of Pain
Keywords: children; nurse; fear; pain; skin prick test
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): Hand puppet was used in the skin prick test process from the children in the experimental group.
  Interventions: Other: Hand puppet method
- Active comprator (Active Comparator): Kaleidoscope was used in the skin prick test process from the children in the experimental group.
  Interventions: Other: Kaleidoscope method
- control group (No Intervention): Routine application of the unit will be made

INTERVENTIONS:
Other: Hand puppet method — Children in the experimental group were shown a hand puppet to distract them during the skin test for allergy.
  Arms: experimental group
Other: Kaleidoscope method — Children in the other experimental group were look at kaleidoscope to distract them during the skin test for allergy.
  Arms: Active comprator

SUMMARY:
This study aimed to determine the effects of hand puppets and kaleidoscopes on some emotional parameters in preschool children who underwent skin prick testing at the pediatric allergy and immunology outpatient clinic.The study was conducted with children aged 3-6 years who underwent skin prick testing for allergy testing.In the study, the Introductory Characteristics of Children and Their Families Form, Wong-Baker Faces Pain Rating Scale (FACES) and Child Fear Scale (CFS) were used to store data.The data were uploaded to the computer and coded by the researchers, and the data were evaluated in the SPSS package program. Sociodemographic data of the children participating in the study are given as numbers and percentage distributions. The data were analyzed according to normal distribution and appropriate tests were used. The statistical significance level of the research was determined as p<0.05. In addition, at the end of the study, with a sufficient sample size, working status was tested with post-hoc power analysis.

DETAILED DESCRIPTION:
Type of Research: It is a randomized controlled type research. Place and Characteristics of the Research: It was conducted in the pediatric allergy and immunology outpatient clinic of Fırat University Hospital, with children aged 3-6 years who underwent skin testing for allergy. Children are accompanied by a companion during their examinations. In the routine, no distraction method is used for children during the procedure.

Allocation into groups was done using simple random sampling. Collection of data Study data were collected in 3 groups. Hand puppet group: The hand puppet was used to divert the attention of the children in the group during the skin prick test. The cost of the hand puppet was covered by the researcher.

Kaleidoscope group: It was used to divert the attention of the children in the kaleidoscope group during the skin prick test. Kaleidoscope, also known as a kaleidoscope, is a play tool that multiplies the outside image when viewed inside. The cost of the kaleidoscope was covered by the researcher.

Control group: No intervention was made to the children in the control group during the skin prick test.

1. In the first stage, randomization of children who met the research criteria was performed.
2. The "Introductory Characteristics Form for Children and Their Families" was filled in for the children assigned to the groups.
3. After the children's doctor's examination at the pediatric allergy and immunology outpatient clinic, the child and his/her family, for whom a skin prick test was requested, were evaluated in the room where the test would be performed. The children in the hand puppet group were started to play games with the hand puppet by the researcher 1 minute before the procedure. During the procedure, the children in the kaleidoscope group were asked to look inside the kaleidoscope and describe the shapes they saw, thus drawing their attention to the shapes in the kaleidoscope. No application was made to the children in the control group during the skin prick test. Children, their families and the observer were asked to answer the "Wong-Baker Faces Pain Rating Scale (FACES)" and "Child Fear Scale (CFS)" questions before and after the treatment. Skin prick test was applied to all children in the sample group by the same nurse, in accordance with the procedure steps.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-6 years.
* The child and his/her parents volunteer to participate in the research.
* No mental or neurological disability,
* Not having a life-threatening disease,
* Children's cognitive level and motor development are appropriate,
* No visual or auditory problems,
* Children who have not undergone any invasive procedure other than skin prick testing.
* Those who have not had a skin prick test before.
* The child does not complain of acute pain. (Pain scale VAS score is 0)

Exclusion Criteria:

* Children requiring intravenous or intramuscular intervention before skin prick test
* Development of complications during the procedure
* Being so agitated that it is impossible to communicate with the child.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
WONG-BAKER FACES PAIN RATING SCALE | day 1
  In this scale, faces are given pain scores according to numerical values. The lowest score is "0" and the highest score is "10". As the score from the scale increases, the intensity of pain increases, and as the score decreases, the intensity decreases.

SECONDARY OUTCOMES:
Children's Fear Scale | day 1
  5 cartoon face pictures were used in the scale. Anxiety level is evaluated with numbers between "0" and "4". A score of "0" indicates "no anxiety" and a score of "4" indicates "severe anxiety".

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem Selime Merter, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tufekci FG, Celebioglu A, Kucukoglu S. Turkish children loved distraction: using kaleidoscope to reduce perceived pain during venipuncture. J Clin Nurs. 2009 Aug;18(15):2180-6. doi: 10.1111/j.1365-2702.2008.02775.x. PMID 19583650
- [Background] Bekar P, Erkul M, Efe E. The effect of using a kaleidoscope during central venous catheter dressing changes on pain and anxiety in children with cancer: A randomised controlled trial. Eur J Oncol Nurs. 2022 Apr;57:102114. doi: 10.1016/j.ejon.2022.102114. Epub 2022 Feb 25. PMID 35248915
- [Background] Semerci R, Akgun Kostak M. The Efficacy of Distraction Cards and Kaleidoscope for Reducing Pain During Phlebotomy: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Aug;35(4):397-402. doi: 10.1016/j.jopan.2020.02.003. Epub 2020 Apr 28. PMID 32354466
- [Background] Bulut M, Kucuk Alemdar D, Bulut A, Salci G. The Effect of Music Therapy, Hand Massage, and Kaleidoscope Usage on Postoperative Nausea and Vomiting, Pain, Fear, and Stress in Children: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Dec;35(6):649-657. doi: 10.1016/j.jopan.2020.03.013. Epub 2020 Jul 20. PMID 32703758
- [Background] Oluc T, Sarialioglu A. The effect of a hand puppet-based therapeutic play for preschool children on the fear and pain associated with blood collection procedure. J Pediatr Nurs. 2023 Sep-Oct;72:e80-e86. doi: 10.1016/j.pedn.2023.06.012. Epub 2023 Jun 15. PMID 37330277